CLINICAL TRIAL: NCT04536805
Title: Relapse in Previously Irradiated Prostate Bed : a Phase I/II Study of Stereotactic Ablative Reirradiation Potentiated by Metformin
Brief Title: Relapse in Previously Irradiated Prostate Bed : Stereotactic Ablative Reirradiation Potentiated by Metformin
Acronym: REPAIR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2020-01
Record Dates: First submitted 2020-08-17; First posted 2020-09-03 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Stereotactic Body Radiation Therapy; SBRT; Metformin; Previously Irradiated Prostate Bed; Biochemical recurrence
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin + SBRT at total dose of 30 Gray (Gy) (Experimental): Metformin: 850 mg per day (day -15 to day 0) 1700 mg per day (day 1 to day 75)
  Stereotactic Body Radiation Therapy (SBRT): Dose escalation 5 x 6 Gy, (day 0 to day 10)
  Interventions: Drug: Metformin; Radiation: Stereotactic Body Radiation Therapy (SBRT) 30 Gray (Gy)
- Metformin + SBRT at total dose of 36 Gy (Experimental): Metformin: 850 mg per day (day -15 to day 0) 1700 mg per day (day 1 to day 75)
  Stereotactic Body Radiation Therapy (SBRT): Dose escalation 6 x 6 Gy (day 0 to day 12)
  Interventions: Drug: Metformin; Radiation: Stereotactic Body Radiation Therapy (SBRT) 36 Gy
- Metformin + SBRT at total dose of 25 Gy (Experimental): Metformin: 850 mg per day (day -15 to day 0) 1700 mg per day (day 1 to day 75)
  Stereotactic Body Radiation Therapy (SBRT): Dose escalation 5 x 5 Gy (day 0 to day 10)
  Interventions: Drug: Metformin; Radiation: Stereotactic Body Radiation Therapy (SBRT) 25 Gy

INTERVENTIONS:
Drug: Metformin — Metformin: 850 mg per day (day -15 to day 0) 1700 mg per day (day 1 to day 75)
Radiation: Stereotactic Body Radiation Therapy (SBRT) 30 Gray (Gy) — Stereotactic Body Radiation Therapy (SBRT): Dose escalation 5 x 6 Gy day 0 to day 10
  Other Names: SBRT
  Arms: Metformin + SBRT at total dose of 30 Gray (Gy)
Radiation: Stereotactic Body Radiation Therapy (SBRT) 36 Gy — Stereotactic Body Radiation Therapy (SBRT): Dose escalation 6 x 6 Gy day 0 to day 12
  Other Names: SBRT
  Arms: Metformin + SBRT at total dose of 36 Gy
Radiation: Stereotactic Body Radiation Therapy (SBRT) 25 Gy — Stereotactic Body Radiation Therapy (SBRT): Dose escalation 5x 5 Gy day 0 to day 10
  Arms: Metformin + SBRT at total dose of 25 Gy

SUMMARY:
This phase I/II escalation dose study is assessing the efficacy of the recommended dose of stereotactic re-irradiation (SBRT) of relapses within the prostatectomy bed, potentiated by metformin

DETAILED DESCRIPTION:
The purpose of this escalation study is, first to select the recommended dose of re-irradiation SBRT in combination with Metformin (based on treatment toxicity monitoring) and then to estimate the efficacy of re-irradiation SBRT in combination with Metformin.

Five or six fractions, at a level of 5 or 6 Gray (Gy) per session (either 5 x 6 Gy, 6 x 6 Gy, or 5 x 5 Gy), will be delivered over a maximum of 12 days (from day 1 to day 10 or 12) to provide a total dose of 25 to 36 Gy.

Patient receive oral Metformin treatment from Day -15 and Day 75.

Patient will be followed for 5 years: patients visits will be planned at week 2; 4; 8; 12; and month M6; M9; M12; M18; M24; M36; 4 years and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to International Conference on Harmonisation (ICH)/ Good Clinical Practice (GCP) regulations before registration and prior to any trial specific procedures.
* Biochemical recurrence occurring at least 2 years after external radiotherapy to the prostate lodge and the end of hormone therapy, for prostatic adenocarcinoma previously treated by radical prostatectomy.
* Local recurrence in irradiated areas proven by biological (PSA > 0.2 ng/ml and ascending confirmed by at least 2 successive assays) and radiological (lesion visible on MRI and/or Choline PET and/or Prostate-Specific Membrane Antigen (PSMA) PET).
* Recurrence without rectal invasion
* Pelvic and prostate MRI evaluation
* Absence of pelvic lymph node or metastatic recurrence proven by choline PET or PSMA PET scan
* World Health Organisation (WHO) performance status 0-1
* Low risk, intermediate risk and high risk with a single risk factor
* PSA doubling time > 6 months
* No anti-cancer treatments planned for the current relapse, including hormone therapy.
* Age > 18 years old.
* Life expectancy greater than or equal to 5 years.
* Patient registered with a health insurance system.
* Patients willing and able to comply with the planned visits, treatment plan, laboratory tests and other study procedures indicated in the protocol.

Exclusion Criteria:

* Metastatic disease (bone, lymph node or other)
* Late radiotherapy urinary or gastrointestinal toxicity (grade ≥ 2) (after radiotherapy of prostate lodge)
* History of cancer in the 5 years prior to trial entry other than cutaneous basal cell carcinoma
* Inflammatory bowel disease
* Contraindications for performing MRI
* Rectal surgery history
* Patient treated for Diabetes
* Creatinine clearance < 45 mL/min
* Treatment with metformin in the last 3 months prior to inclusion
* Severe comorbidity that may affect treatment, for example :

  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of inclusion.
  * Unstable angina, myocardial infarction and/or congestive heart failure requiring hospitalization within the last 6 months
  * Myocardial infarction in the last 6 months.
  * Exacerbation of Chronic Obstructive Pulmonary Disease (COPD) or other respiratory conditions requiring hospitalization or preventing metformin therapy at the time of inclusion.
* Any condition associated with an increased risk of lactic acidosis (e.g., alcohol abuse, New York Heart Association (NYHA) III or IV congestive heart failure).
* Clinically significant history of hepatopathy with Child-Pugh B or C score, including viral infection or hepatitis, alcohol abuse or cirrhosis.
* Any acute or chronic condition that may result in tissue hypoxia (e.g. heart or respiratory failure, shock).
* Bilateral hip prosthesis
* Treatment with any investigational drug or participation in a clinical trial within 30 days prior to inclusion.
* Known hypersensitivity to metformin or any of its components
* Inability or reluctance to swallow oral medications
* Persons deprived of liberty, under a measure of safeguard of justice, under guardianship or under the tutor authority
* Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Enrollment: 44 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
For phase 1:. Select the recommended dose for SBRT (either 5 x 6 Gy, 6 x 6 Gy, or 5 x 5 Gy), in combination with Metformin | 12 weeks
  SBRT toxicity will be reported during the 12 weeks following the initiation of SBRT.
For phase 2: estimate the efficacy of re-irradiation SBRT in combination with Metformin in terms of biochemical relapse-free survival rate. | 3 years
  PSA levels will be assessed every 3 months within 3 years after SBRT.

SECONDARY OUTCOMES:
Estimate the efficacy of re-irradiation SBRT in combination with Metformin in terms of biochemical relapse-free survival and biochemical response | 5 years
  PSA levels will be assessed every 3 months within 5 years after SBRT.
  For all patients, visits will be made at 6, 9, 12, 18, 24, 36 months, 4 years, and 5 years will be made from the start of SBRT. The end of the trial is defined by the last visit of the last included patient.
Estimation of the efficacy of SBRT re-irradiation in combination with Metformin in terms of progression-free survival and overall survival | 5 years
  Clinical progression-free survival is defined as the time interval between the date of SBRT start and the date of clinical progression (local progression assessed by the physical examination, or appearance of metastatic lesions), start of hormonal therapy or death irrespective of the cause.
Evaluation of acute and late genitourinary and gastrointestinal toxicities of the SBRT re-irradiation | 5 years
  Acute and late genitourinary toxicities over the first 5 years will be assessed according to the NCI-CTCAE V5.0 classification
Evaluation of Quality of life after SBRT re-irradiation in combination with Metformin | 5 years
  Quality of life will be assessed based on EORTC Quality of life questionnaire (QLQ)-C30 scale at week 4; 8; 12; and month M6; M9; M12; M18; M24; M36; 4 years and 5 years. The Time Until Definitive Deterioration (TUDD) will be computed from registration until the first observation of a definitive deterioration of the quality of life, defined as a score decreased by 10 points (in the case of global health scale and functional scales) or increased by 10 points (in the case of symptom scales) compared to the score at baseline, without later improvement superior to 10 points compared to baseline score.
Evaluation of Quality of life after SBRT re-irradiation in combination with Metformin | 5 years
  Quality of life will be assessed based on EORTC Quality of life questionnaire in prostate cancer (QLQ-PR25) scale at week 4; 8; 12; and month M6; M9; M12; M18; M24; M36; 4 years and 5 years. The Time Until Definitive Deterioration (TUDD) will be computed from registration until the first observation of a definitive deterioration of the quality of life, defined as a score decreased by 10 points (in the case of global health scale and functional scales) or increased by 10 points (in the case of symptom scales) compared to the score at baseline, without later improvement superior to 10 points compared to baseline score.
Evaluation of urinary symptoms | 5 years
  Urinary symptoms over the first 5 years will be assessed by International Prostatic Symptom Score (IPSS). This score evaluates the severity of prostate symptoms in the last month on a scale of 0 to 35 (total of 7 items rated 0 to 5).The distributions of this score will be described at inclusion, at follow-up visits (M6 M9 M12 M18 M24 M36 4 and 5 years) and at the end of the study visit according to the following categories:
  0 - 7: Poorly symptomatic ; 8 - 19: Moderately symptomatic ; 20 - 35: Severe symptoms.
Evaluation of erectile function | 5 years
  Erectile function will be assessed by International Index of Erectile Function (IIEF5). This score assesses erectile function over the past 6 months on a scale of 1 to 25 (total of 5 items rated 0/1 to 5). The distributions of this score will be described at baseline, at follow-up visits (M6 M12 M18, M24,M36 4 and 5 years old) and at the end of the study visit according to the following categories:
  1 - 4: Non-interpretable ; 5 - 10: Severe erectile dysfunction ; 11 - 15: Moderate erectile dysfunction ; 16 - 20: Mild erectile dysfunction ; 21 - 25: Normal erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: Valentine GUIMAS, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (12):
- France (12):
  - Institut de Cancerologie de L'Ouest, Angers
  - CHRU de BREST - HOPITAL MORVAN, Brest
  - Societe de Recherche Oncologique Clinique 37 (Roc 37), Chambray-lès-Tours
  - Centre GEORGES FRANCOIS LECLERC, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre OSCAR LAMBRET, Lille
  - Centre LEON BERARD, Lyon
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Chru Bretonneau, Tours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary study manuscript after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months and ending 3 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal not overlapping with any planned secondary publications from the research team will be able to access the IPD. To achieve aims in the approved proposal. Proposals should be directed to Chief Investigator who will discuss such requested with the Department of Clinical Research and Innovation (DRCI):
  Valentine.guimas@ico.unicancer.fr. To gain access, data requesters will need to sign a data access agreement. Data will be available for 3 years at Institut de Cancérologie de l'Ouest.

REFERENCES:
- [Derived] Joly A, Blanc Lapierre A, Rio E, Vaugier L, Supiot S, Guimas V. REPAIR_GETUG P16 relapse in previously irradiated prostate bed: a phase I/II study of stereotactic ablative reirradiation potentiated by a metformine study protocol. BMJ Open. 2025 Jul 24;15(7):e100031. doi: 10.1136/bmjopen-2025-100031. PMID 40707156